CLINICAL TRIAL: NCT04012021
Title: EXplanted LIver and Ex-vivo Pancreatic Specimen Evaluation by 7 TESLA MRI - The EXLIPSE Study
Brief Title: EXplanted LIver and Ex-vivo Pancreatic Specimen Evaluation by 7 TESLA MRI
Acronym: EXLIPSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other); Imago 7 (Other)
Responsible Party: Principal Investigator, Laura Crocetti, Associate Professor, University of Pisa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13646
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Liver Cirrhosis; Liver Steatosis; Hepatocellular Carcinoma; Pancreatic Cancer; Magnetic Resonance Imaging
Keywords: liver; cirrhosis; steatosis; hepatocellular carcinoma; pancreatic cancer; 7 tesla; magnetic resonance imaging
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver; Carcinoma, Hepatocellular; Pancreatic Neoplasms; Fibrosis

STUDY DESIGN:
Intervention Model Description: Three single groups to be included
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EX-VIVO SPECIMENS (Experimental): Three groups of ex-vivo surgical specimen:
  Group A: native livers in transplant recipients Group B: liver grafts excluded for donation Group C: primary pancreatic cancer
  Interventions: Diagnostic Test: 7T Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: 7T Magnetic Resonance Imaging — * T1-weighted and T2-weighted sequences
  * quantitative magnetic resonance imaging approach
  * proton spectrum analyses

SUMMARY:
Aim of this study is to evaluate the correlation between the characteristics detected by the 7T MRI equipment and the histological composition of native explanted livers (group A), liver graft excluded for donation (group B) and surgical specimens of primary pancreatic tumour, which underwent pancreaticoduodenectomy (group C).

ELIGIBILITY:
GROUP A of Native Liver

Inclusion Criteria:

* informed consent
* full possession of one's faculties
* patients who are going to undergo liver transplantation, independently from previous therapy or from the primary disease they are affected by.

Exclusion Criteria:

* patients affected by polycystic liver disease
* excluded from liver transplantation.

GROUP B of Excluded Grafts

Inclusion Criteria:

- liver grafts with histologically proven macrovescic steatosis, not fit for transplantation

Exclusion Criteria:

* liver grafts histologically proven macrovescic steatosis fit for transplantation
* liver grafts not fit for transplantation due to causes other than steatosis

GROUP C of Focal Pancreatic Lesion

Inclusion Criteria:

* informed consent
* full possession of one's faculties
* pancreatic lesion assessed by CT examination and histologically proved, which are candidates for pancreaticoduodenectomy or total pancreatectomy

Exclusion Criteria:

- excluded from surgery due to the severity of their condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-24 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the correlation between the characteristics detected by the MRI equipment and the histological composition of ex-vivo specimens from hepatic and pancreatic tissues and lesions | 3 years
  The creation of a data-bank will increase the knowledge about imaging features able to characterize many diseases affecting the liver, and to evaluate cell changes that occur in pancreatic cancer and the tumour pathways of spreading; moreover it will provide a reference framework to define proper acquisition protocols for future clinical applications.
  Such data will also provide imaging biomarkers of malignant cells, and show the morphological changes that occur in neoplastic lesions after systemic or loco-regional therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Crocetti, MD,PhD, Principal Investigator — University of Pisa
Locations (1):
- Azienda Ospedaliero Universitaria Pisana, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kraff O, Fischer A, Nagel AM, Monninghoff C, Ladd ME. MRI at 7 Tesla and above: demonstrated and potential capabilities. J Magn Reson Imaging. 2015 Jan;41(1):13-33. doi: 10.1002/jmri.24573. Epub 2014 Jan 30. PMID 24478137
- [Background] Pohmann R, Speck O, Scheffler K. Signal-to-noise ratio and MR tissue parameters in human brain imaging at 3, 7, and 9.4 tesla using current receive coil arrays. Magn Reson Med. 2016 Feb;75(2):801-9. doi: 10.1002/mrm.25677. Epub 2015 Mar 29. PMID 25820458
- [Background] Stephenson MC, Gunner F, Napolitano A, Greenhaff PL, Macdonald IA, Saeed N, Vennart W, Francis ST, Morris PG. Applications of multi-nuclear magnetic resonance spectroscopy at 7T. World J Radiol. 2011 Apr 28;3(4):105-13. doi: 10.4329/wjr.v3.i4.105. PMID 21532871
- [Background] Terpstra M, Cheong I, Lyu T, Deelchand DK, Emir UE, Bednarik P, Eberly LE, Oz G. Test-retest reproducibility of neurochemical profiles with short-echo, single-voxel MR spectroscopy at 3T and 7T. Magn Reson Med. 2016 Oct;76(4):1083-91. doi: 10.1002/mrm.26022. Epub 2015 Oct 26. PMID 26502373
- [Background] Zakhari S. Bermuda Triangle for the liver: alcohol, obesity, and viral hepatitis. J Gastroenterol Hepatol. 2013 Aug;28 Suppl 1:18-25. doi: 10.1111/jgh.12207. PMID 23855291
- [Background] Meyers RL, Tiao GM, Dunn SP, McGahren ED 3rd, Langham MR Jr; Central Surgical Review Committee, Children's Oncology Group AHEP-0731, Treatment of Children with All Stages Hepatoblastoma. Surgical management of children with locally advanced hepatoblastoma. Cancer. 2012 Aug 15;118(16):4090-1; author reply 4094-5. doi: 10.1002/cncr.26715. Epub 2012 Jul 3. No abstract available. PMID 22760520
- [Background] Grossman EJ, Millis JM. Liver transplantation for non-hepatocellular carcinoma malignancy: Indications, limitations, and analysis of the current literature. Liver Transpl. 2010 Aug;16(8):930-42. doi: 10.1002/lt.22106. PMID 20677284
- [Background] Dhir M, Lyden ER, Smith LM, Are C. Comparison of outcomes of transplantation and resection in patients with early hepatocellular carcinoma: a meta-analysis. HPB (Oxford). 2012 Sep;14(9):635-45. doi: 10.1111/j.1477-2574.2012.00500.x. Epub 2012 Jun 19. PMID 22882201
- [Background] Lim KB, Schiano TD. Long-term outcome after liver transplantation. Mt Sinai J Med. 2012 Mar-Apr;79(2):169-89. doi: 10.1002/msj.21302. PMID 22499489
- [Background] Yao FY. Liver transplantation for hepatocellular carcinoma: beyond the Milan criteria. Am J Transplant. 2008 Oct;8(10):1982-9. doi: 10.1111/j.1600-6143.2008.02351.x. Epub 2008 Aug 22. PMID 18727702
- [Background] Yao FY, Bass NM, Nikolai B, Davern TJ, Kerlan R, Wu V, Ascher NL, Roberts JP. Liver transplantation for hepatocellular carcinoma: analysis of survival according to the intention-to-treat principle and dropout from the waiting list. Liver Transpl. 2002 Oct;8(10):873-83. doi: 10.1053/jlts.2002.34923. PMID 12360427
- [Background] Sposito C, Droz Dit Busset M, Citterio D, Bongini M, Mazzaferro V. The place of liver transplantation in the treatment of hepatic metastases from neuroendocrine tumors: Pros and cons. Rev Endocr Metab Disord. 2017 Dec;18(4):473-483. doi: 10.1007/s11154-017-9439-7. PMID 29359266
- [Background] Nakao A, Harada A, Nonami T, Kaneko T, Takagi H. Clinical significance of carcinoma invasion of the extrapancreatic nerve plexus in pancreatic cancer. Pancreas. 1996 May;12(4):357-61. doi: 10.1097/00006676-199605000-00006. PMID 8740402
- [Background] Lehmann A, Denkert C, Budczies J, Buckendahl AC, Darb-Esfahani S, Noske A, Muller BM, Bahra M, Neuhaus P, Dietel M, Kristiansen G, Weichert W. High class I HDAC activity and expression are associated with RelA/p65 activation in pancreatic cancer in vitro and in vivo. BMC Cancer. 2009 Nov 13;9:395. doi: 10.1186/1471-2407-9-395. PMID 19912635
- [Background] Loos M, Hedderich DM, Ottenhausen M, Giese NA, Laschinger M, Esposito I, Kleeff J, Friess H. Expression of the costimulatory molecule B7-H3 is associated with prolonged survival in human pancreatic cancer. BMC Cancer. 2009 Dec 26;9:463. doi: 10.1186/1471-2407-9-463. PMID 20035626
- [Background] Shepherd TM, Thelwall PE, Stanisz GJ, Blackband SJ. Aldehyde fixative solutions alter the water relaxation and diffusion properties of nervous tissue. Magn Reson Med. 2009 Jul;62(1):26-34. doi: 10.1002/mrm.21977. PMID 19353660
- [Background] Yong-Hing CJ, Obenaus A, Stryker R, Tong K, Sarty GE. Magnetic resonance imaging and mathematical modeling of progressive formalin fixation of the human brain. Magn Reson Med. 2005 Aug;54(2):324-32. doi: 10.1002/mrm.20578. PMID 16032673